CLINICAL TRIAL: NCT03090152
Title: Minimal Opioid Use After Total Hip Replacement (THR): a Blinded Randomized Placebo-controlled Study
Brief Title: Minimal Opioid Use After Total Hip Replacement (THR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-0721
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Replacement; Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Periarticular Injection (PAI) (Active Comparator): * Aspirin and nerve pain medications including duloxetine and clonidine patch prior to surgery.
  * Peri-articular injection in the operating room
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * A pain regimen while in the hospital that includes EPCA (saline) Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Interventions: Procedure: Periarticular injection (Deep injection); Procedure: Periarticular injection (Superficial injection); Drug: Placebo
- Epidural Patient-Controlled Analg (EPCA) (Active Comparator): * Aspirin and nerve pain medications including duloxetine and clonidine patch prior to surgery.
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * A pain regimen while in the hospital that consists of Epidural PCA (EPCA) with 0.06% bupivacaine. Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV The EPCA will be removed when pain is well-controlled. Other medications, including opioids, will be available.
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Interventions: Drug: Bupivacaine
- PAI + EPCA (Experimental): * Aspirin and nerve pain medications including duloxetine and clonidine
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * Anesthetic, Antiemetic and peri-articular injection in the operating room
  * A pain regimen while in the hospital that consists of EPCA (with 0.06% bupivacaine) Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV The EPCA will be removed when pain is well-controlled. Other medications, including opioids, will be available.
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Interventions: Procedure: Periarticular injection (Deep injection); Procedure: Periarticular injection (Superficial injection); Drug: Bupivacaine

INTERVENTIONS:
Procedure: Periarticular injection (Deep injection) — Deep injection of "cocktail" containing Bupivacaine with Epi, 30mL; Morphine, 8mg/mL, 1mL; Methyprednislone, 40mg/mL, 1mL; Cefazolin, 500mg in 10 mL; saline, 22mL into the anterior capsule, the periosteum, the gluteus maximus, and the abductor muscles and fascia lata.
  Arms: PAI + EPCA; Periarticular Injection (PAI)
Procedure: Periarticular injection (Superficial injection) — Superficial injection of 40mL 0.25% Bupivacaine into subcutaneous tissue prior to wound closure.
  Arms: PAI + EPCA; Periarticular Injection (PAI)
Drug: Bupivacaine — EPCA: Bupivacaine 0.06%.
  Arms: Epidural Patient-Controlled Analg (EPCA); PAI + EPCA
Drug: Placebo — EPCA: Saline.
  Arms: Periarticular Injection (PAI)

SUMMARY:
Total hip arthroplasty can be associated with significant postoperative pain. Side effects of pain management may impair participation in physical therapy and slow readiness for discharge from the hospital. In a previous study done by the investigators' group, epidural patient controlled analgesia (EPCA) with a hydromorphone containing solution appeared to have a more favorable pain profile with ambulation, but greater side effects compared to injection of a peri-articular cocktail. The use of opioid was greater in the peri-articular injection group (PAI). There was no difference in length of stay. In view of the controversy over opioid use, the investigators would like to develop an optimal opioid sparing pain management approach by comparing 3 different protocols 1) Plain local anesthetic EPCA; 2) PAI; 3) EPCA + PAI; all in conjunction with a multimodal opioid sparing pain regimen. The goal would be to maximize pain control while minimizing opioid use and side-effects.

DETAILED DESCRIPTION:
Long acting narcotics or scheduled doses of narcotics are often used as part of a multimodal pain regimen. In this study, this is eliminated. Instead, it uses a cocktail of different drugs including intraoperative Ketamine use (NMDA receptor antagonist), intra-op Benadryl (to decrease excitation of nociceptors) and IV Tylenol. The narcotic free regimen starts preoperatively with the use of Aspirin,Clonidine patch, Cymbalta (Duloxetine), and is maintained both intraoperatively and post operatively. Baby ASA (81mg) is being used as an anti-inflammatory agent. A number of studies including the one by Morris et al. (2009), have shown via in vitro experiments that low dose aspirin decreases polymorphonuclear leukocyte and macrophage accumulation. It inhibits thromboxane making it an antithrombotic agent as well. The concern with aspirin has been major bleeding. Several studies in the orthopedic patient population using ≤81 mg of aspirin have shown that it does not increase bleeding (Cuellar, Mantz). At HSS, patients are routinely continued on baby aspirin when needed for its cardio protective effect. Devereaux in the POISE trial did show an increased risk of bleeding when ASA was given preoperatively at a dose of 200 mg. In our study, all patients will be given intravenous tranexamic acid which should mitigate against the risk of bleeding. Duloxetine is also being added. In a recent study done at HSS. Duloxetine was found to decrease the amount of opioid use and nausea. If found to be more effective with the use of EPCA vs. PAI or combination of the two, a new way of managing postop pain while minimizing Nnartcuoreti co fu Ssetu adsy per CDC recommendation will be helpful in managing patients post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with osteoarthritis scheduled for primary total hip arthroplasty with a participating surgeon
* Planned use of regional anesthesia
* Planned posterolateral surgical approach
* Age Range 45-80
* Ability to follow study protocol

Exclusion Criteria:

* Any patient with age <45 or >80
* Any patient with planned anterior surgical approach
* Any patient with prior major ipsilateral hip surgery
* Any patient intending to receive general anesthesia
* Any patient with an ASA of IV
* Any patient with insulin-dependent diabetes
* Any patient with hepatic (liver) failure (history of cirrhosis or elevated LFT's)
* Any patient with chronic renal (kidney) failure (formal diagnosis of renal disease of elevated creatinine)
* Any patient with history of gastric (stomach) ulcer
* Chronic opioid use (taking opioids for >3 mo duration on a daily basis)
* Chronic analgesic use (i.e. lyrica, gabapentin) for >3 mo duration
* Stress dose steroids
* Use of antidepressants
* Contraindications to aspirin
* Allergy to any of the medications (or adhesives) involved in the study protocol
* Dementia
* Non-English speakers.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy Jules-Elysee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Periarticular Injection (PAI): * Aspirin and nerve pain medications including duloxetine and clonidine patch prior to surgery.
  * Peri-articular injection in the operating room
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * A pain regimen while in the hospital that includes EPCA (saline) Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Periarticular injection (Deep injection): Deep injection of "cocktail" containing Bupivacaine with Epi, 30mL; Morphine, 8mg/mL, 1mL; Methyprednislone, 40mg/mL, 1mL; Cefazolin, 500mg in 10 mL; saline, 22mL into the anterior capsule, the periosteum, the gluteus maximus, and the abductor muscles and fascia lata.
  Periarticular injection (Superficial injection): Superficial injection of 40mL 0.25% Bupivacaine into subcutaneous tissue prior to wound closure.
  Placebo: EPCA: Saline.
- Epidural Patient-Controlled Analg (EPCA): * Aspirin and nerve pain medications including duloxetine and clonidine patch prior to surgery.
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * A pain regimen while in the hospital that consists of Epidural PCA (EPCA) with 0.06% bupivacaine. Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV The EPCA will be removed when pain is well-controlled. Other medications, including opioids, will be available.
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Bupivacaine: EPCA: Bupivacaine 0.06%.
- PAI + EPCA: * Aspirin and nerve pain medications including duloxetine and clonidine
  * Combined Spinal Epidural with 1.5% Mepivacaine 4cc
  * Anesthetic, Antiemetic and peri-articular injection in the operating room
  * A pain regimen while in the hospital that consists of EPCA (with 0.06% bupivacaine) Duloxetine (Cymbalta) - by mouth Ketorolac (Toradol) - IV Celecoxib (Celebrex) - by mouth Acetaminophen (Tylenol) - IV The EPCA will be removed when pain is well-controlled. Other medications, including opioids, will be available.
  * Acetaminophen and celecoxib for pain control once out of the hospital. Patients will also receive a prescription for an opioid medication in case they need it.
  Periarticular injection (Deep injection): Deep injection of "cocktail" containing Bupivacaine with Epi, 30mL; Morphine, 8mg/mL, 1mL; Methyprednislone, 40mg/mL, 1mL; Cefazolin, 500mg in 10 mL; saline, 22mL into the anterior capsule, the periosteum, the gluteus maximus, and the abductor muscles and fascia lata.
  Periarticular injection (Superficial injection): Superficial injection of 40mL 0.25% Bupivacaine into subcutaneous tissue prior to wound closure.
  Bupivacaine: EPCA: Bupivacaine 0.06%.
Period: Overall Study
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Started | 60 | 60 | 60
Completed | 59 | 56 | 59
Not Completed | 1 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Surgery Canceled | 1 | 0 | 0
Not completed — Epidural catheter could not be placed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA | Total
Number analyzed (Participants) | 59 | 56 | 59 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8) | 64 (7) | 64 (7) | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 32 | 84
  Male | 30 | 33 | 27 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 2 | 9
  Not Hispanic or Latino | 54 | 54 | 57 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 6
  White | 54 | 53 | 56 | 163
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 59 | 56 | 59 | 174

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: Oral morphine equivalents, cumulative
Time Frame: within 24 hours after surgery
Measure: Mean (Inter-Quartile Range); unit: Oral Morphine Equivalent (mg)
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
Oral Morphine Equivalent (mg) | 30 [15 to 45] | 22.5 [7.5 to 45] | 15 [7.5 to 30]

2. Secondary Outcome: Pain at Rest
Description: NRS (Numeric Pain Rating Scale). 0 means no pain, 10 means worst pain imaginable. A lower score is a better outcome.
Time Frame: Postoperative Day 1,2,3,7,90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
score on a scale
  POD1 | 2 (1.9) | 1.9 (1.8) | 1.7 (1.8)
  POD2 | 2.2 (2) | 1.8 (1.9) | 1.9 (1.8)
  POD3 | 1.8 (1.6) | 1.2 (1.5) | 1.3 (1.4)
  POD7 | 1.5 (1.8) | 1.1 (1.4) | 1.5 (1.7)
  POD90 | 0.3 (0.8) | 0.3 (0.7) | 0.6 (1.3)

3. Secondary Outcome: Pain With Activity
Description: NRS (Numeric Pain Rating Scale). 0 means no pain, 10 means worst pain imaginable. A lower score is a better outcome.
Time Frame: Postoperative Day 1,2,3,7,90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
score on a scale
  POD1 | 3.6 (2.4) | 3.4 (2.3) | 3.7 (2.6)
  POD2 | 4.2 (2.3) | 3.6 (2.5) | 4 (2.1)
  POD3 | 3.8 (2.5) | 3.2 (2.2) | 3.2 (2.1)
  POD7 | 2.8 (2.1) | 2.7 (1.9) | 3 (2)
  POD90 | 0.7 (1.2) | 0.6 (1.2) | 1.4 (2.1)

4. Secondary Outcome: Opioid Side Effects
Description: via ORSDS (Opioid-Related Symptom Distress Scale). Each symptom was rated on a 4 point scale from 0-4. A lower score is a better outcome.
Time Frame: Postoperative Day 1,2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
score on a scale
  POD1- Fatigue | 0.8 (1.2) | 0.6 (0.9) | 0.9 (1.1)
  POD1- Drowsiness | 1.1 (1) | 0.6 (0.9) | 1.3 (1.1)
  POD1- Inability to Concentrate | 0.2 (0.6) | 0.1 (0.5) | 0.3 (0.8)
  POD1- Nausea | 0.7 (1.2) | 0.3 (0.7) | 0.6 (1)
  POD1- Dizziness | 0.4 (0.7) | 0.5 (1) | 0.9 (1)
  POD1- Constipation | 0.2 (0.6) | 0.5 (1) | 0.4 (0.8)
  POD2- Fatigue | 0.7 (1) | 0.7 (1.1) | 1 (1.2)
  POD2- Drowsiness | 1 (1) | 0.7 (1) | 1.2 (1.1)
  POD2- Inability to Concentrate | 0.2 (0.6) | 0.1 (0.4) | 0.3 (0.8)
  POD2- Nausea | 0.2 (0.6) | 0.3 (0.9) | 0.6 (1.1)
  POD2-Dizziness | 0.4 (0.8) | 0.4 (0.9) | 0.6 (1.1)
  POD2- Constipation | 0.7 (1.1) | 0.7 (1.1) | 1 (1.3)

5. Secondary Outcome: Patient Satisfaction
Description: via Likert scale. A higher score is a better outcome. the scale is from 0-10.
Time Frame: Postoperative Day 1,2,3,7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
score on a scale
  POD1 | 9.6 (1.3) | 9.6 (0.8) | 9.5 (1.1)
  POD2 | 9.3 (1.5) | 9.1 (1.5) | 9.1 (1.2)
  POD3 | 9.5 (1) | 9.1 (1.5) | 9.1 (1.4)
  POD7 | 9.6 (0.9) | 9.4 (0.8) | 8.9 (2.2)

6. Secondary Outcome: Post-operative Pain
Description: via PAINOUT (Improvement in postoperative PAIN OUTcome) Minumum value is zero, maximum is ten. Higher scores mean worse outcomes.
Time Frame: Postoperative Day 1
Population: some patients were lost to follow up or did not answer questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 58 | 55 | 56
score on a scale
  The worst pain you had in the last 24 hours | 5.5 [2 to 7] | 5 [3 to 7] | 4 [2 to 7]
  The least pain you had in the last 24 hours | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
  How often were you in severe pain in the last 24 hours? | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
  How much pain interfered with doing activities in bed like turning, sitting up, changing position? | 1 [0 to 3] | 2 [0 to 5] | 1 [0 to 3]
  How much pain interfered with or prevented you from breathing deeply or coughing? | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  How much pain interfered with or prevented you from sleeping? | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  How much pain interfered with doing activities out of bed? | 2 [0 to 4] | 2 [0 to 5] | 2 [0 to 4]
  In the last 24 hours, have you had any nausea? | 0 [0 to 4] | 0 [0 to 0] | 0 [0 to 3]
  In the last 24 hours, have you had any drowsiness? | 2.5 [0 to 5] | 0 [0 to 3] | 3 [0 to 5]
  In the last 24 hours, have you had any itching? | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Neuropathic Pain Assessed With S-LANSS
Description: via S-LANSS (Self-report Leeds Assessment of Neuropathic Symptoms and Signs). Scores range from 0-24. A lower score is a better outcome.
Time Frame: Postoperative Day 7, Postoperative Day 90
Population: some patients were Lost to Follow up or did not answer questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 58
score on a scale
  POD7: number analyzed (Participants) | 48 | 47 | 50
  POD7 | 8 [5 to 8] | 8 [5 to 8] | 7.5 [5 to 8]
  POD90: number analyzed (Participants) | 45 | 36 | 36
  POD90 | 8 [8 to 8] | 8 [8 to 8] | 8 [8 to 8]

8. Secondary Outcome: Quality of Recovery
Description: Via QoR-40 (Quality of Recovery). Minimum value of 40, maximum of 200. Higher values mean better outcome
Time Frame: Postoperative Day 1,2,3
Population: Lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 58 | 54 | 58
score on a scale
  POD1 | 102.2 (6.6) | 102.3 (5.9) | 101.6 (6.8)
  POD2: number analyzed (Participants) | 54 | 51 | 57
  POD2 | 102.9 (7.4) | 103.1 (7.4) | 102.1 (7.8)
  POD3: number analyzed (Participants) | 52 | 53 | 54
  POD3 | 100.7 (7) | 98.5 (8.9) | 98.4 (8.8)

9. Secondary Outcome: Readiness for Discharge Time
Description: When patient meets all readiness for discharge criteria
Time Frame: From end of surgery until the date/time of first documented clearance for discharge, assessed up to 1 week.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 58 | 56 | 59
hours | 46.5 [27.8 to 49.9] | 48.7 [30.7 to 51.1] | 48.8 [43.9 to 51.2]

10. Secondary Outcome: Blinding Assessment
Description: What group do you think you were in
Time Frame: Assessed on day of discharge and on seventh post operative day
Population: Lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 50 | 52 | 51
Participants
  Discharge: PAI | 5 | 13 | 7
  Discharge: EPCA | 10 | 10 | 6
  Discharge: PAI+EPCA | 18 | 11 | 15
  Discharge: Do Not Know | 17 | 18 | 23
  POD7: number analyzed (Participants) | 46 | 45 | 42
  POD7: PAI | 6 | 8 | 7
  POD7: EPCA | 6 | 3 | 4
  POD7: PAI+EPCA | 17 | 16 | 13
  POD7: Do Not Know | 17 | 18 | 18

11. Secondary Outcome: Opioid Consumption During the First 3 Days Post-op
Description: Opioids consumed in the first 3 after surgery (cumulative consumption).
Time Frame: Postoperative day 0,1,2,3
Measure: Median (Inter-Quartile Range); unit: Oral Morphine Equivalent (mg)
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
Oral Morphine Equivalent (mg) | 52.5 [22.5 to 105] | 45 [15 to 105] | 40 [15 to 85]

12. Secondary Outcome: No Opioids Consumed
Description: Number of patients who did not consume any opioids
Time Frame: 0 to 24 hours post-operatively
Measure: Number; unit: participants
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
Number analyzed (Participants) | 59 | 56 | 59
participants | 5 | 12 | 14

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Periarticular Injection (PAI) | Epidural Patient-Controlled Analg (EPCA) | PAI + EPCA
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03090152/Prot_SAP_000.pdf